CLINICAL TRIAL: NCT02581267
Title: Missed Serious Medical Illness in Psychiatric Patients Seen in an Academic Emergency Department
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: Western University, Canada (Other)
Responsible Party: Principal Investigator, Chris Poss, Resident, Western University, Canada
Other Study IDs: 107073
Record Dates: First submitted 2015-08-08; First posted 2015-10-20 (Estimated); Last update posted 2015-10-20 (Estimated); Status verified 2015-10

CONDITIONS: Emergency Services, Psychiatric

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective

SUMMARY:
Psychiatric presentations are common in the emergency department (ED), and determining whether or not a psychiatric presentation is due to medical illness can be a difficult task for the emergency physician. The investigators define "serious medical illness" (SMI) as a pathological condition that would necessitate inpatient treatment on a medical or surgical ward. It is important for patient safety that SMI be triaged by the emergency physician to the appropriate inpatient service. The rate of missed SMI in patients with psychiatric presentations to the ED is unknown. The investigators will research missed SMI in patients referred to adult psychiatry from the ED, with the intent to improve patient safety.

ELIGIBILITY:
Inclusion Criteria:

* All patients greater than or equal to 18 years of age presenting to London Health Sciences Centre, Victoria Hospital emergency department between October 1, 2014 - July 31, 2015 who were referred to adult psychiatry by the emergency physician.

Exclusion Criteria:

* None

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adults emergency room patients referred to adult psychiatry by the emergency physician
Sampling Method: Non-Probability Sample
Enrollment: 800 (Estimated)
Dates: Start 2015-10; Primary Completion 2015-12 (Estimated); Study Completion 2015-12 (Estimated)

PRIMARY OUTCOMES:
Number of patients admitted to a medical / surgical service within 7 days of psychiatry referral in the emergency department | Approximately 8 months
Medical / surgical admission diagnosis | Approximately 8 months
  This will be extracted from the electronic medial record.
Number of days after psychiatric referral that patient is admitted to medical / surgical service | Approximately 8 months

SECONDARY OUTCOMES:
Proportion of patients discharged home from the emergency department by psychiatry following referral by the emergency physician | Approximately 8 months
Risk factors associated with medical / surgical admission after initial psychiatry referral | Approximately 8 months
  The investigators will be extracting variables from the patient's chart including triage vital signs, past medical and psychiatric history, initial laboratory bloodwork, and determining if any of these are risk factors for subsequent medical / surgical admission.
Number of admissions to medical / surgical service within 30 days of discharge from psychiatry | Approximately 8 months